CLINICAL TRIAL: NCT02954419
Title: IgA Nephropathy Biomarkers Evaluation Study (INTEREST)
Acronym: INTEREST
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: SYSU-PRGIgAN-003
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: IgA Nephropathy; Glomerular Diseases
Keywords: IgA Nephropathy; Biomarker
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples of the patients are collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IgA nephropathy group: Eligible biopsy-proven primary IgA nephropathy patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This prospective cohort study is designed to examine the association between blood and urine biomarkers (including genetic variants) and long-term kidney disease progression among 2000 Chinese IgA nephropathy patients with relatively normal kidney function (eGFR≥60 ml/min/1.73 m2).

DETAILED DESCRIPTION:
Glomerulonephritis is the leading cause of end-stage renal disease (ESRD) in China, where IgA nephropathy (IgAN) is the most common primary glomerulonephritis among individuals undergoing renal biopsy. The outcomes of IgAN vary highly among individuals; some have the stable renal function for lifetime and some quickly progress to ESRD. No biomarker is widely applied to predict the outcomes in IgAN yet. Previous GWAS studies including ours have identified some susceptibility loci associated with the development and clinical features of IgAN. In addition, a few cohort studies have revealed several genetic loci related to the progression of IgAN. But, all of the reported GWAS studies were based on a case-control design, which may not provide the information about the effect of genetic variants on the progression of disease. Previous cohort studies which focused on certain specific candidate genes cannot unbiasedly explore the progression related susceptibility loci. Furthermore, there is no study that integrates the information from whole genomic loci and serum and urine biomarkers to predict the long-term progression in IgAN. Therefore, we design a relative large prospective cohort study to examine the association between blood and urine biomarkers (including whole genomic loci) and long-term kidney disease progression among 2000 Chinese IgAN patients with relatively normal kidney function (eGFR≥60 ml/min/1.73 m2).

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals aged 14 years or older
* Patients with biopsy-proven primary IgA nephropathy
* A renal biopsy available for reviewing must include 10 or more glomeruli.
* The first renal biopsy was performed within 3 years.
* eGFR ≥ 60 ml/min/1.73 m2 (MDRD formula);
* Individuals or their legal representative who are able to understand and have voluntarily signed the informed consent form (ICF).

Exclusion Criteria:

* Relatives were diagnosed with biopsy-proven primary IgA nephropathy;
* Individuals had secondary IgA nephropathy due to diseases such as diabetes, chronic liver disease and systemic lupus erythematosus.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with biopsy-proven primary IgA nephropathy
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
A doubling of serum creatinine level from baseline | 120 months
Progression to end stage renal disease (eGFR<15ml/min/1.73 m2, dialysis or transplantation） | 120 months
Death | 120 months

SECONDARY OUTCOMES:
Remission of proteinuria (complete or partial) | 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Xue Qing Yu, M.D. & Ph.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided